CLINICAL TRIAL: NCT04617834
Title: Enhancing Rural Health Via Cardiovascular Telehealth for Rural Patients (E-VICTORS) Project
Brief Title: Enhancing Rural Health Via Cardiovascular Telehealth for Rural Patients Implementation (E-VICTORS)
Acronym: E-VICTORS
Status: Active, not recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB00068612
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Acute Coronary Syndrome
Keywords: acute chest pain; telehealth; implementation science; rural health
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality Surveillance Data: For this quality surveillance study, data will be collected retrospectively through electronic health record (EHR) queries for all eligible patients treated for acute cardiovascular symptoms by one of the study sites.
  Interventions: Other: Quality Surveillance Data Collection

INTERVENTIONS:
Other: Quality Surveillance Data Collection — Data will be retrospectively collected through EHR queries

SUMMARY:
This pre-post study will evaluate the implementation of a cardiovascular telehealth platform, which will connect experts from the Wake Forest University Health Sciences (WFUHS) tertiary care center with Wilkes County Emergency Medical Services (WC-EMS) system, Wilkes Medical Center Emergency Department (ED), and The Wilkes County Health Department Public Health Community Clinic (PHCC) to improve cardiovascular care in this rural community.

DETAILED DESCRIPTION:
This program aims to improve cardiovascular care for patients in Wilkes County by implementing a cardiovascular telehealth program designed to; a) assist WC- EMS paramedics with the early risk stratification (electrocardiogram (EKG) interpretation, vital signs, and risk scores), treatment, and transportation destination decisions in patients with acute chest pain or dyspnea, b) support Wilkes Medical Center (WMC) Emergency Department (ED) providers (physicians and advanced practice clinicians) in the evaluation, management, and disposition of patients with acute cardiovascular symptoms, and c) provide consultative expertise to the Primary Health Care Centers (PHCC) for patients seen following an EMS or ED encounter for cardiovascular symptoms.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years at time of index encounter
* Cardiovascular symptoms (chest discomfort or dyspnea consistent with possible ACS) as indicated by the treating provider

Exclusion Criteria:

* Age <18
* Traumatic chest pain
* Dyspnea that is clearly from a non-cardiac etiology
* Patients with hemodynamic instability SBP < 90 mmHg, HR>160 or <40 bpm
* Patients requiring intubation/mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is adult patients with cardiovascular symptoms. Therefore, adult patients (>18 years old) with acute chest pain or dyspnea concerning for acute cardiovascular disease will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Emergency Department (ED) utilization | baseline
  ED utilization among patients with cardiovascular symptoms will be defined as the total number of cardiovascular-related ED admissions divided by the total number of unique individual patients receiving cardiovascular care during the project period.

SECONDARY OUTCOMES:
Number of Cardiovascular hospitalizations | Baseline
  Cardiovascular hospitalizations will be defined as an inpatient or observation admission for cardiovascular conditions or symptoms based on Current Procedures Terminology (CPT) and International Classification of Diseases (ICD) codes
Number of Cardiovascular Inter-facility transfers | Baseline
  Cardiovascular Inter-facility transfers will be defined based on patients with cardiovascular symptoms or conditions transferred from Wilkes Medical Center (WMC) to another hospital.
Number of 30-day cardiovascular Emergency Department (ED) re-admissions | day 30
  30-day cardiovascular ED re-admissions will be defined as any cardiovascular related ED admission occurring during the 30 days following their initial/index ED encounter.
Number of 30-day cardiovascular hospital re-admissions | day 30
  30-day cardiovascular hospital re-admissions will be defined as any cardiovascular related hospital admission occurring during the 30 days following their index hospitalization.
Number of Adverse Events | day 30 and Month 12
  Determine if telehealth implementation will result in improved sorting of cases for escalated and de-escalated care, reducing the number of adverse events.
Change in Cost - societal level | day 30 and Month 12
  Evaluate whether spending on healthcare (i.e., insurance payments) changes during the 30-day follow-up period.
Change in Cost - provider level | day 30 and Month 12
  Estimates will be obtained for the impact of the establishment of the telehealth program on the budget of the tertiary center.
Cost-effectiveness | Month 12 and Month 48
  Cost-effectiveness: will be evaluated at the societal level to inform the relative changes in patient outcomes and costs resulting from the telehealth program.
Cardiovascular telehealth consultation rate | Baseline
  Cardiovascular telehealth consultation rate will be assessed by identifying the total number of patients that received cardiovascular telehealth consultations at each originating site divided by the total number of patients at each originating site with cardiovascular symptoms.
Cardiovascular telehealth adoption rate | Month 12
  Adoption rate will be defined by the cardiovascular telehealth consultation rate at each originating site during the first 12 months following implementation of the cardiovascular telehealth service.
Cardiovascular telehealth sustainability rate | Month 24 - Month 48 post Intervention
  Sustainability rate will be defined by the cardiovascular telehealth consultation rate at each site greater than 12 months after the availability of the cardiovascular telehealth service.

OTHER OUTCOMES:
(ED) Emergency Department length of stay (LOS) | Baseline
  ED LOS will be defined as the time from the patient's ED arrival to ED discharge, transfer, or admission
Time to transfer | Baseline
  Time to transfer will be defined by the time between a physician order for transfer and the patient leaving the ED
Patient satisfaction Score | Day 30 and year 1
  Patient satisfaction will be measured (telephone follow-ups) using a modified Short Assessment of Patient Satisfaction (SAPS) which is a validated 7 question instrument, which uses a 5-point Likert scale - scoring: 0 to 10 = Very dissatisfied; 11 to 18 = Dissatisfied; 19 to 26 = Satisfied; 27 to 28 = Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Simon A Mahler, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - Wilkes County Emergency Medical Services, Wilkesboro, North Carolina
  - Wilkes County Public Health Community Clinic, Wilkesboro, North Carolina
  - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Stafford R, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):948-54. doi: 10.1161/CIRCULATIONAHA.109.192666. No abstract available. PMID 20177011
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):143-52. doi: 10.1161/CIR.0b013e318282ab8f. No abstract available. PMID 23283859
- [Background] Jollis JG, Al-Khalidi HR, Roettig ML, Berger PB, Corbett CC, Doerfler SM, Fordyce CB, Henry TD, Hollowell L, Magdon-Ismail Z, Kochar A, McCarthy JJ, Monk L, O'Brien P, Rea TD, Shavadia J, Tamis-Holland J, Wilson BH, Ziada KM, Granger CB. Impact of Regionalization of ST-Segment-Elevation Myocardial Infarction Care on Treatment Times and Outcomes for Emergency Medical Services-Transported Patients Presenting to Hospitals With Percutaneous Coronary Intervention: Mission: Lifeline Accelerator-2. Circulation. 2018 Jan 23;137(4):376-387. doi: 10.1161/CIRCULATIONAHA.117.032446. Epub 2017 Nov 14. PMID 29138292
- [Background] Abrams TE, Vaughan-Sarrazin M, Kaboli PJ. Mortality and revascularization following admission for acute myocardial infarction: implication for rural veterans. J Rural Health. 2010 Fall;26(4):310-7. doi: 10.1111/j.1748-0361.2010.00318.x. Epub 2010 Aug 17. PMID 21029165
- [Background] Lambert L, Brown K, Segal E, Brophy J, Rodes-Cabau J, Bogaty P. Association between timeliness of reperfusion therapy and clinical outcomes in ST-elevation myocardial infarction. JAMA. 2010 Jun 2;303(21):2148-55. doi: 10.1001/jama.2010.712. PMID 20516415
- [Background] James CV, Moonesinghe R, Wilson-Frederick SM, Hall JE, Penman-Aguilar A, Bouye K. Racial/Ethnic Health Disparities Among Rural Adults-United States, 2012-2015: MMWR Surveillance Summaries / November 17, 2017 / 66(23);1-9. J Health Care Poor Underserved. 2018;29(1):19-34. doi: 10.1353/hpu.2018.0003. PMID 29503284
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines: developed in collaboration with the American College of Emergency Physicians and Society for Cardiovascular Angiography and Interventions. Catheter Cardiovasc Interv. 2013 Jul 1;82(1):E1-27. doi: 10.1002/ccd.24776. Epub 2013 Jan 8. No abstract available. PMID 23299937
- [Background] Harrington RA, Califf RM, Balamurugan A, Brown N, Benjamin RM, Braund WE, Hipp J, Konig M, Sanchez E, Joynt Maddox KE. Call to Action: Rural Health: A Presidential Advisory From the American Heart Association and American Stroke Association. Circulation. 2020 Mar 10;141(10):e615-e644. doi: 10.1161/CIR.0000000000000753. Epub 2020 Feb 10. PMID 32078375
- [Background] Mahler SA, Hiestand BC, Goff DC Jr, Hoekstra JW, Miller CD. Can the HEART score safely reduce stress testing and cardiac imaging in patients at low risk for major adverse cardiac events? Crit Pathw Cardiol. 2011 Sep;10(3):128-33. doi: 10.1097/HPC.0b013e3182315a85. PMID 21989033
- [Background] Mahler SA, Riley RF, Hiestand BC, Russell GB, Hoekstra JW, Lefebvre CW, Nicks BA, Cline DM, Askew KL, Elliott SB, Herrington DM, Burke GL, Miller CD. The HEART Pathway randomized trial: identifying emergency department patients with acute chest pain for early discharge. Circ Cardiovasc Qual Outcomes. 2015 Mar;8(2):195-203. doi: 10.1161/CIRCOUTCOMES.114.001384. Epub 2015 Mar 3. PMID 25737484
- [Background] Mahler SA, Lenoir KM, Wells BJ, Burke GL, Duncan PW, Case LD, Herrington DM, Diaz-Garelli JF, Futrell WM, Hiestand BC, Miller CD. Safely Identifying Emergency Department Patients With Acute Chest Pain for Early Discharge. Circulation. 2018 Nov 27;138(22):2456-2468. doi: 10.1161/CIRCULATIONAHA.118.036528. PMID 30571347
- [Background] Stopyra JP, Riley RF, Hiestand BC, Russell GB, Hoekstra JW, Lefebvre CW, Nicks BA, Cline DM, Askew KL, Elliott SB, Herrington DM, Burke GL, Miller CD, Mahler SA. The HEART Pathway Randomized Controlled Trial One-year Outcomes. Acad Emerg Med. 2019 Jan;26(1):41-50. doi: 10.1111/acem.13504. Epub 2018 Jul 19. PMID 29920834
- [Background] Stopyra JP, Harper WS, Higgins TJ, Prokesova JV, Winslow JE, Nelson RD, Alson RL, Davis CA, Russell GB, Miller CD, Mahler SA. Prehospital Modified HEART Score Predictive of 30-Day Adverse Cardiac Events. Prehosp Disaster Med. 2018 Feb;33(1):58-62. doi: 10.1017/S1049023X17007154. Epub 2018 Jan 10. PMID 29316995
- [Background] Stopyra JP, Snavely AC, Scheidler JF, Smith LM, Nelson RD, Winslow JE, Pomper GJ, Ashburn NP, Hendley NW, Riley RF, Koehler LE, Miller CD, Mahler SA. Point-of-Care Troponin Testing during Ambulance Transport to Detect Acute Myocardial Infarction. Prehosp Emerg Care. 2020 Nov-Dec;24(6):751-759. doi: 10.1080/10903127.2020.1721740. Epub 2020 Mar 3. PMID 31985326
- [Background] Proctor EK, Powell BJ, McMillen JC. Implementation strategies: recommendations for specifying and reporting. Implement Sci. 2013 Dec 1;8:139. doi: 10.1186/1748-5908-8-139. PMID 24289295
- [Background] Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. Implement Sci. 2015 Feb 12;10:21. doi: 10.1186/s13012-015-0209-1. PMID 25889199
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Gesell SB, Golden SL, Limkakeng AT Jr, Carr CM, Matuskowitz A, Smith LM, Mahler SA. Implementation of the HEART Pathway: Using the Consolidated Framework for Implementation Research. Crit Pathw Cardiol. 2018 Dec;17(4):191-200. doi: 10.1097/HPC.0000000000000154. PMID 30418249
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Erhardt L, Herlitz J, Bossaert L, Halinen M, Keltai M, Koster R, Marcassa C, Quinn T, van Weert H; Task Force on the management of chest pain. Task force on the management of chest pain. Eur Heart J. 2002 Aug;23(15):1153-76. doi: 10.1053/euhj.2002.3194. No abstract available. PMID 12206127
- [Background] Kerr D, Holden D, Smith J, Kelly AM, Bunker S. Predictors of ambulance use in patients with acute myocardial infarction in Australia. Emerg Med J. 2006 Dec;23(12):948-52. doi: 10.1136/emj.2006.038414. PMID 17130609
- [Background] Larson DM, Menssen KM, Sharkey SW, Duval S, Schwartz RS, Harris J, Meland JT, Unger BT, Henry TD. "False-positive" cardiac catheterization laboratory activation among patients with suspected ST-segment elevation myocardial infarction. JAMA. 2007 Dec 19;298(23):2754-60. doi: 10.1001/jama.298.23.2754. PMID 18165668
- [Background] Brunetti ND, Dellegrottaglie G, Lopriore C, Di Giuseppe G, De Gennaro L, Lanzone S, Di Biase M. Prehospital telemedicine electrocardiogram triage for a regional public emergency medical service: is it worth it? A preliminary cost analysis. Clin Cardiol. 2014 Mar;37(3):140-5. doi: 10.1002/clc.22234. Epub 2014 Jan 22. PMID 24452666
- [Background] Langabeer JR 2nd, Champagne-Langabeer T, Alqusairi D, Kim J, Jackson A, Persse D, Gonzalez M. Cost-benefit analysis of telehealth in pre-hospital care. J Telemed Telecare. 2017 Sep;23(8):747-751. doi: 10.1177/1357633X16680541. Epub 2016 Dec 5. PMID 27913657
- [Background] Mohr NM, Young T, Harland KK, Skow B, Wittrock A, Bell A, Ward MM. Emergency Department Telemedicine Shortens Rural Time-To-Provider and Emergency Department Transfer Times. Telemed J E Health. 2018 Aug;24(8):582-593. doi: 10.1089/tmj.2017.0262. Epub 2018 Jan 2. PMID 29293413
- [Background] Stopyra J, Snavely AC, Hiestand B, Wells BJ, Lenoir KM, Herrington D, Hendley N, Ashburn NP, Miller CD, Mahler SA. Comparison of accelerated diagnostic pathways for acute chest pain risk stratification. Heart. 2020 Jul;106(13):977-984. doi: 10.1136/heartjnl-2019-316426. Epub 2020 Apr 8. PMID 32269131
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Psaty BM, Delaney JA, Arnold AM, Curtis LH, Fitzpatrick AL, Heckbert SR, McKnight B, Ives D, Gottdiener JS, Kuller LH, Longstreth WT Jr. Study of Cardiovascular Health Outcomes in the Era of Claims Data: The Cardiovascular Health Study. Circulation. 2016 Jan 12;133(2):156-64. doi: 10.1161/CIRCULATIONAHA.115.018610. Epub 2015 Nov 4. PMID 26538580
- [Background] Hawthorne G, Sansoni J, Hayes L, Marosszeky N, Sansoni E. Measuring patient satisfaction with health care treatment using the Short Assessment of Patient Satisfaction measure delivered superior and robust satisfaction estimates. J Clin Epidemiol. 2014 May;67(5):527-37. doi: 10.1016/j.jclinepi.2013.12.010. PMID 24698296
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Chit A, Becker DL, DiazGranados CA, Maschio M, Yau E, Drummond M. Cost-effectiveness of high-dose versus standard-dose inactivated influenza vaccine in adults aged 65 years and older: an economic evaluation of data from a randomised controlled trial. Lancet Infect Dis. 2015 Dec;15(12):1459-66. doi: 10.1016/S1473-3099(15)00249-2. Epub 2015 Sep 8. PMID 26362172
- [Background] Dauerman HL, Bates ER, Kontos MC, Li S, Garvey JL, Henry TD, Manoukian SV, Roe MT. Nationwide Analysis of Patients With ST-Segment-Elevation Myocardial Infarction Transferred for Primary Percutaneous Intervention: Findings From the American Heart Association Mission: Lifeline Program. Circ Cardiovasc Interv. 2015 May;8(5):e002450. doi: 10.1161/CIRCINTERVENTIONS.114.002450. PMID 25901044
- [Background] Langabeer JR 2nd, Prasad S, Seo M, Smith DT, Segrest W, Owan T, Gerard D, Eisenhauer MD. The effect of interhospital transfers, emergency medical services, and distance on ischemic time in a rural ST-elevation myocardial infarction system of care. Am J Emerg Med. 2015 Jul;33(7):913-6. doi: 10.1016/j.ajem.2015.04.009. Epub 2015 Apr 10. PMID 25910668
- [Background] Rhudy JP Jr, Alexandrov AW, Hyrkas KE, Jablonski-Jaudon RA, Pryor ER, Wang HE, Bakitas MA. Geographic access to interventional cardiology services in one rural state. Heart Lung. 2016 Sep-Oct;45(5):434-40. doi: 10.1016/j.hrtlng.2016.07.002. Epub 2016 Aug 1. PMID 27493022
- [Background] Tanguay A, Dallaire R, Hebert D, Begin F, Fleet R. Rural Patient Access to Primary Percutaneous Coronary Intervention Centers is Improved by a Novel Integrated Telemedicine Prehospital System. J Emerg Med. 2015 Nov;49(5):657-64. doi: 10.1016/j.jemermed.2015.05.009. Epub 2015 Jul 26. PMID 26215451
- [Background] American College of Emergency Physicians Clinical Policies Subcommittee (Writing Committee) on Suspected Non-ST-Elevation Acute Coronary Syndromes:; Tomaszewski CA, Nestler D, Shah KH, Sudhir A, Brown MD. Clinical Policy: Critical Issues in the Evaluation and Management of Emergency Department Patients With Suspected Non-ST-Elevation Acute Coronary Syndromes. Ann Emerg Med. 2018 Nov;72(5):e65-e106. doi: 10.1016/j.annemergmed.2018.07.045. PMID 30342745
- See also: CMS Rural Health Strategy, Accessed 8/27/2018 — https://www.cms.gov/About-CMS/Agency-Information/OMH/Downloads/Rural-Strategy-2018.pdf
- See also: Bureau USC. United States Census Bureau QuickFacts. 2020 — https://www.census.gov/quickfacts/NC
- See also: Access NC Community Demographics Search. Accessed May 12, 2020. — https://accessnc.nccommerce.com/DemographicsReports/
- See also: HPSA Find — https://data.hrsa.gov/tools/shortage-area/hpsa-find
- See also: MUA Find — https://data.hrsa.gov/tools/shortage-area/mua-find
- See also: Quality AfHRa. Medical Expenditure Panel Survey. Bethesda, MA2020. — https://www.meps.ahrq.gov/mepsweb/
- See also: Medicare Fee-For-Service Payment — https://www.cms.gov/Regulations-and-Guidance/Regulations-and-Policies/Medicare-Fee-for-Service-Payment-Regulations
- See also: Health Insurance Coverage in the United States: 2018: United States Census Bureau — https://www.census.gov/library/publications/2019/demo/p60-267.html
- See also: Bureau USC. American Community Survey (ACS). — https://www.census.gov/programs-surveys/acs
- See also: Bureau USC. Type of Health Insurance Coverage by State: 2013, 2017, and 2018. — https://www.census.gov/library/visualizations/interactive/health-insurance-coverage-type.html
- See also: Local Area Unemployment Statistics Information and Analysis — https://data.bls.gov/lausmap/showMap.jsp;jsessionid=3BD90BDBDF311A4CFBC957F639625EE5._t3_07v